CLINICAL TRIAL: NCT00849680
Title: A Phase I Dose-Ranging Study of the Safety, Tolerability, and Immunogenicity of the Merck Trivalent Adenovirus Serotype 5 HIV-1 Gag/Pol/Nef Vaccine (MRKAd5 HIV-1 Gag/Pol/Nef) in a Prime-Boost Regimen in Healthy Adults
Brief Title: A Study of Safety, Tolerability, and Immunogenicity of the MRKAd5 Gag/Pol/Nef Vaccine in Healthy Adults (V520-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V520-016; 2009_548
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: HIV-1; HIV Infections
Keywords: HIV Seronegativity; Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo (Placebo Comparator): Participants receiving 1.0 ml of placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine or the placebo to the MRKAd5 HIV-1 gag vaccine injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26 or a 2-dose regimen at Day 1 and Week 26 or Day 1 and Week 4.
  Interventions: Other: Comparator: Placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine; Biological: Comparator: Placebo to MRKAd5 HIV-1 gag vaccine
- Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose) (Experimental): Participants receiving 1.0 ml of the Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26.
  Interventions: Biological: Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose)
- Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose) (Experimental): Participants receiving 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26.
  Interventions: Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose)
- Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose) (Experimental): Participants receiving 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26.
  Interventions: Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose)
- Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose) (Experimental): Participants receiving 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26.
  Interventions: Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose)
- Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose) (Experimental): Participants receiving 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26.
  Interventions: Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose)
- Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose) (Experimental): Participants receiving 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26, or in a 2-dose regimen at Day 1 and Week 4 (with no vaccine administered at Week 26) or Day 1 and Week 26 (with placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine administered at Week 4)
  Interventions: Other: Comparator: Placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine; Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose)
- Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose) (Experimental): Participants receiving 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose) injected intramuscularly in a 3-dose regimen at Day 1, Week 4 and Week 26.
  Interventions: Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose)

INTERVENTIONS:
Other: Comparator: Placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine — Placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine.
  Arms: Placebo; Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose)
Biological: Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose) — Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose)
  Other Names: V520
  Arms: Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose)
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose)
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose)
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose)
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose)
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose)
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose)
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose)
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose)
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose)
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose)
Biological: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose) — Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose)
  Other Names: V520
  Arms: Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose)
Biological: Comparator: Placebo to MRKAd5 HIV-1 gag vaccine — Placebo to the MRKAd5 HIV-1 gag vaccine.
  Arms: Placebo

SUMMARY:
The goal of this study is to understand the safety, tolerability and immunogenicity of the Merck Trivalent Adenovirus Serotype 5 HIV-1 gag/pol/nef

Vaccine (MRKAd 5 HIV-1 gag/pol/nef) vaccine in healthy human volunteers compared to placebo. The study will also evaluate a number of dose levels and the necessity for and timing of booster injections.

DETAILED DESCRIPTION:
The study will proceed in four stages. Following stages I, II and III, all subjects will have the Postdose 1 (PD1) clinical and laboratory safety data reviewed by the Safety Evaluation Committee (SEC). If these data are acceptable, the next stage will be initiated.

* In Stage I, participants will be randomized to receive 3 doses of the 3x10^9vp/dose level Trivalent vaccine or placebo.
* In Stage II, participants will be randomized to receive 2 or 3 doses of the 3x10^10vp/dose level Trivalent vaccine or placebo.
* In Stage III, participants will be randomized to receive 3 doses of the Trivalent vaccine with titers of 1x10^11vp/dose, 3x10^6vp/dose, 3x10^7vp/dose, or 3x10^8vp/dose or placebo.
* In Stage IV, participants will be randomized to all treatment groups. In addition, some participants will be randomized to an MRKAd 5 HIV-1 gag Monovalent vaccine. In this stage, participants will be pre-stratified by baseline Ad5 titers (=<200, and >200), to ensure an even distribution of participants with high and low Ad5 titers across the various treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 Years to 45 Years in Stages I-III and 18 Years to 50 Years in Stage IV.
* Subject is in good general health
* Subjects of reproductive potential agree to use acceptable method of birth control through study
* Subject tests negative for Hepatitis B, Hepatitis C, and HIV

Exclusion Criteria:

* Subject has a recent history of fever at time of vaccination
* Subject has received immune globulin or blood product 3 months prior to injection
* Subject has been vaccinated with live virus vaccine 30 days prior to receipt of first dose
* Subject has been vaccinated with inactivated vaccine with 14 days prior to receipt of first dose
* Subject has a chronic medical condition that is considered progressive
* Subject has history of malignancy
* Subject weighs less than 105 lb.
* Female subject is pregnant or breast feeding, Male subject is planning to impregnate during the first year of study
* Subject has contraindication to intramuscular injection
* Subject has a tattoo on the deltoid region of the arm or the injection of Depo-Provera
* Subject is unlikely or unwilling to adhere to lower risk sex practices during the course of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2003-04; Primary Completion 2005-03 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Priddy FH, Brown D, Kublin J, Monahan K, Wright DP, Lalezari J, Santiago S, Marmor M, Lally M, Novak RM, Brown SJ, Kulkarni P, Dubey SA, Kierstead LS, Casimiro DR, Mogg R, DiNubile MJ, Shiver JW, Leavitt RY, Robertson MN, Mehrotra DV, Quirk E; Merck V520-016 Study Group. Safety and immunogenicity of a replication-incompetent adenovirus type 5 HIV-1 clade B gag/pol/nef vaccine in healthy adults. Clin Infect Dis. 2008 Jun 1;46(11):1769-81. doi: 10.1086/587993. PMID 18433307
- [Derived] Li F, Finnefrock AC, Dubey SA, Korber BT, Szinger J, Cole S, McElrath MJ, Shiver JW, Casimiro DR, Corey L, Self SG. Mapping HIV-1 vaccine induced T-cell responses: bias towards less-conserved regions and potential impact on vaccine efficacy in the Step study. PLoS One. 2011;6(6):e20479. doi: 10.1371/journal.pone.0020479. Epub 2011 Jun 10. PMID 21695251
- [Derived] Hutnick NA, Carnathan DG, Dubey SA, Cox KS, Kierstead L, Makadonas G, Ratcliffe SJ, Lasaro MO, Robertson MN, Casimiro DR, Ertl HC, Betts MR. Vaccination with Ad5 vectors expands Ad5-specific CD8 T cells without altering memory phenotype or functionality. PLoS One. 2010 Dec 22;5(12):e14385. doi: 10.1371/journal.pone.0014385. PMID 21203546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 317 participants were randomized. 2 did not receive any study medication. Therefore, the safety population was 315.
Groups:
- Placebo: 2 or 3 doses of 1.0 mg of placebo to the MRKAd5 HIV-1 gag/pol/nef vaccine or 3 doses of placebo to the MRKAd5 HIV-1 gag vaccine injected intramuscularly.
- Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose): 3 doses of 1.0 ml of the Monovalent MRKAd5 HIV-1 gag vaccine (1x10^9 vp/dose) injected intramuscularly.
- Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose): 3 doses of 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^6 vp/dose) injected intramuscularly.
- Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose): 3 doses of 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^7 vp/dose) injected intramuscularly.
- Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose): 3 doses of 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^8 vp/dose) injected intramuscularly.
- Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose): 3 doses of 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^9 vp/dose) injected intramuscularly.
- Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose): 2 or 3 doses of 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (3x10^10 vp/dose) injected intramuscularly.
- Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose): 3 doses of 1.0 ml of Trivalent MRKAd5 HIV-1 gag/pol/nef vaccine (1x10^11 vp/dose) injected intramuscularly.
Period: Overall Study
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose)
Started | 27 | 13 | 42 | 42 | 42 | 42 | 78 | 31
Completed | 16 | 10 | 27 | 28 | 32 | 27 | 61 | 23
Not Completed | 11 | 3 | 15 | 14 | 10 | 15 | 17 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 7 | 3 | 12 | 11 | 8 | 11 | 12 | 5
Not completed — Subject moved | 1 | 0 | 3 | 1 | 0 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 2 | 2 | 1 | 1
Not completed — Subject unable to comply with protocol | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose) | Total
Number analyzed (Participants) | 27 | 13 | 42 | 42 | 42 | 42 | 78 | 31 | 317
Age, Customized [Mean (Full Range); unit: Years] | 32.4 [19 to 50] | 34.3 [18 to 46] | 33.2 [19 to 50] | 32.6 [19 to 50] | 33.3 [18 to 50] | 34.0 [18 to 50] | 35.7 [19 to 50] | 34.8 [19 to 50] | 34.0 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 21 | 14 | 17 | 21 | 31 | 14 | 149
  Male | 8 | 1 | 21 | 28 | 25 | 21 | 47 | 17 | 168
Region of Enrollment [Number; unit: participants]
  United States | 27 | 13 | 42 | 42 | 42 | 42 | 78 | 31 | 317

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Experiences
Description: Adverse experiences (AE) collected include serious and non serious systemic AEs, and injection-site AEs.
  Systemic and Laboratory AEs include any unfavorable & unintended change in the structure, function, or chemistry of the body.
  Injection-site AEs include any swelling, redness, pain or tenderness at the injection site. All injection site AEs were collected up to 5 days after any vaccine dose.
Time Frame: up to 260 weeks after first vaccination
Measure: Number; unit: Participants
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose)
Number analyzed (Participants) | 27 | 13 | 41 | 42 | 42 | 41 | 78 | 31
Participants
  With non-serious systemic AEs (NSAE) | 20 | 13 | 36 | 33 | 35 | 37 | 68 | 28
  With Injection site AEs | 6 | 9 | 17 | 18 | 22 | 23 | 57 | 29
  With serious systemic AEs | 1 | 2 | 2 | 3 | 4 | 3 | 7 | 1
  With serious injection site AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Laboratory Adverse Experiences
Description: Laboratory AEs were based on a grading system considering the severity of abnormal laboratory values in participants and reflect any unfavorable and unintentional change in function, or chemistry of the body.
  All laboratory AEs were collected up to 29 days after any vaccine dose.
Time Frame: up to 260 weeks after first vaccination
Population: Participants administered at least one dose of study vaccine. One participant who was lost to follow-up, and another one participant who discontinued as he comply with the protocol are not included.
Measure: Number; unit: Participants
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose)
Number analyzed (Participants) | 25 | 13 | 41 | 42 | 42 | 41 | 78 | 31
Participants
  With non-serious laboratory AEs | 10 | 5 | 12 | 6 | 12 | 17 | 29 | 11
  With serious laboratory AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Immune Response by Levels of Unfractionated Gag, Pol, and Nef-specific IFN-gamma Following a 3-dose Vaccine Regimen
Description: Participants expressing HIV antigens (gag, pol and nef) secrete antigen specific interferon-gamma (IFN-gamma). Levels of unfractionated gag, pol, and nef-specific IFN-gamma were to be measured using an Enzyme Linked Immunospot Assay (ELISPOT), which measures spot forming cells per 10^6 peripheral blood mononuclear cells (SFC per million PBMCs).
Time Frame: 4 weeks after booster injection
Population: No immunogenicity analyses were performed because the results from a previous study, V520-023 (NCT00095576), which used the same vaccine as the one used in this study (NCT00849680) proved it was not efficacious.
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Immune Response by Levels of Unfractionated Gag, Pol, and Nef-specific IFN-gamma Following a 2-dose Vaccine Regimen
Description: Participants expressing HIV antigens (gag, pol and nef) secrete antigen specific interferon-gamma (IFN-gamma). Levels of unfractionated gag, pol, and nef-specific IFN-gamma were to be measured using an Enzyme Linked Immunospot Assay (ELISPOT), which measures spot forming cells per 10^6 peripheral blood mononuclear cells (SFC per million PBMCs).
  No immunogenicity analyses were performed because the results from a previous study, V520-023 (NCT00095576), which used the same vaccine as the one used in this study (NCT00849680) proved it was not efficacious.
Time Frame: 4 weeks after booster injection
Population: as for outcome 3
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^6 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^7 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^8 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^9 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10^10 vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10^11 vp/Dose)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10[9] vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[6] vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[7] vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[8] vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[9] vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[10] vp/Dose) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10[11] vp/Dose)
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/13 | 2/41 | 3/42 | 4/42 | 3/42 | 7/78 | 1/31
Other Adverse Events (participants affected / at risk) | 24/26 | 13/13 | 35/41 | 38/42 | 35/42 | 39/42 | 74/78 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10[9] vp/Dose) (N=13) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[6] vp/Dose) (N=41) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[7] vp/Dose) (N=42) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[8] vp/Dose) (N=42) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[9] vp/Dose) (N=42) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[10] vp/Dose) (N=78) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10[11] vp/Dose) (N=31)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Monovalent MRKAd5 HIV-1 Gag Vaccine (1x10[9] vp/Dose) (N=13) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[6] vp/Dose) (N=41) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[7] vp/Dose) (N=42) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[8] vp/Dose) (N=42) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[9] vp/Dose) (N=42) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (3x10[10] vp/Dose) (N=78) | Trivalent MRKAd5 HIV-1 Gag/Pol/Nef Vaccine (1x10[11] vp/Dose) (N=31)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (2) | 2 (10) | 1 (1) | 1 (1) | 2 (4)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 3 (3) | 7 (7) | 7 (8) | 5 (6) | 10 (17) | 11 (12) | 7 (11)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 14 (17) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
Chills (General disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 18 (21) | 9 (12)
Fatigue (General disorders) | 3 (3) | 4 (6) | 5 (8) | 7 (10) | 6 (8) | 12 (14) | 20 (23) | 12 (18)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Injection site erythema (General disorders) | 4 (6) | 4 (5) | 6 (6) | 6 (6) | 7 (9) | 8 (10) | 15 (19) | 11 (14)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 5 (9) | 8 (19) | 13 (18) | 13 (20) | 21 (40) | 22 (42) | 56 (114) | 29 (68)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Injection site swelling (General disorders) | 1 (3) | 3 (3) | 0 (0) | 4 (4) | 5 (6) | 8 (9) | 17 (22) | 10 (14)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 2 (4)
Pain (General disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (4) | 0 (0) | 4 (5) | 10 (13) | 4 (5)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (3) | 6 (7) | 5 (7) | 21 (30) | 11 (19)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (4) | 2 (2) | 2 (2) | 2 (2) | 4 (5) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (3) | 4 (4) | 6 (7) | 5 (5) | 4 (5) | 13 (16) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 8 (10) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (5) | 1 (1) | 3 (5) | 1 (1)
Bacteria urine identified (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 2 (4) | 1 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 4 (8) | 4 (8) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 3 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (7) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 2 (2) | 1 (2) | 2 (3) | 2 (2)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 3 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 2 (4) | 2 (2) | 2 (2) | 1 (1)
Red blood cells urine positive (Investigations) | 5 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 8 (16) | 0 (0)
Urinary sediment present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (3)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 4 (7) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 4 (4) | 2 (5) | 3 (3) | 3 (3) | 3 (3) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 4 (4) | 4 (5) | 6 (18) | 3 (4) | 14 (19) | 8 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 12 (24) | 6 (12) | 10 (25) | 13 (17) | 13 (26) | 12 (19) | 35 (69) | 14 (23)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (4) | 4 (7) | 0 (0) | 6 (6) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 5 (5) | 2 (2) | 8 (9) | 6 (6) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 6 (7) | 1 (1) | 10 (12) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (6) | 8 (11) | 5 (5) | 12 (18) | 10 (16) | 13 (16) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
An interim analysis of a related study, V520 Protocol 023 (NCT00095576), showed that the MRKAd5 vaccine used in Protocol 016 (NCT00849680) was not efficacious; therefore, only a high level summary of the safety data was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study is part of a multicenter trial, publications derived from this study should include input from the principal investigator, his/her colleagues, the other investigators in this trial, and SPONSOR personnel.

The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication guidelines.